CLINICAL TRIAL: NCT06178042
Title: Evaluation of the Efficiency of Different Remineralization Methods Used In the Treatment of Post-Orthodontic White Spot Lesions With Quantitative Light-Induced Fluorescence Method
Brief Title: Effectiveness of MI Paste Plus and Remin Pro on Remineralization of Post-Orthodontic White Spot Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, SEVGİ GÖL PEYNİRCİ, Principal investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPEYNIRCI
Record Dates: First submitted 2023-09-18; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: White Spot Lesion; Remineralization
Keywords: White Spot Lesion; Remineralization; QLF; ICDAS II

STUDY DESIGN:
Intervention Model Description: Thirty-nine patients were randomized in a 1:1:1 ratio to either MI Paste Plus or Remin Pro or control group.
Who Masked: Outcomes Assessor
Masking Description: Blinding was not feasible during the intervention, but the data evaluation and outcome assessment were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MI Paste Plus (Experimental): Patients were instructed to use MI Paste Plus (GC Europe, Leuven, Belgium) according to manufacturers instructions.
  Interventions: Combination Product: MI Paste Plus
- Remin Pro (Experimental): Patients were instructed to use (Remin Pro, VOCO GmbH, Cuxhaven, Germany) a pea-sized amount of the cream.
  Interventions: Combination Product: Remin Pro
- Control (Active Comparator): Patients used a 1450 ppm fluoridated tooth paste (Colgate Sensitive Pro-Relief, Colgate-Palmolive, Swidnica, Poland) for conventional tooth brushing.
  Interventions: Combination Product: Control

INTERVENTIONS:
Combination Product: MI Paste Plus — Briefly, a pea-sized amount of the cream was used once a day and was allowed to remain on the teeth for three minutes after conventional tooth brushing. Patient was advised to not to spit out the cream for 30 seconds to activate the product with saliva. Patient was advised to spit out the remaining amount to avoid swallowing excessive fluoride and to wait for 30 minutes after the treatment before rinsing or eating or drinking.
  Arms: MI Paste Plus
Combination Product: Remin Pro — The cream must remain on the teeth for at least three minutes once daily after conventional tooth brushing. Patient was advised to spit out the remaining amount to avoid swallowing excessive fluoride and to wait for 30 minutes after the treatment before rinsing or eating or drinking.
  Arms: Remin Pro
Combination Product: Control — Patients instructed to follow a routine home care.
  Arms: Control

SUMMARY:
One of the most undesired side effects of fixed orthodontic treatment is white spot lesions (WSLs), that appear on the buccal surface of teeth and cause aesthetic problems. The aim of this prospective study was to quantitively evaluate the remineralization effect of casein phosphopeptide-amorphous calcium fluorophosphate (CPP-ACFP) containing (MI Paste Plus®) and hydroxyapatite, xylitol and fluoride containing (Remin Pro®) agents in remineralizing post orthodontics white spots using Quantitive Light-Induced Fluorescence Method (QLF) and ICDAS II criteria, compared to a control group in whom just a routine home care was instructed. Thirty-nine individuals who had recently completed orthodontic treatment, had at least one WSL on upper anterior teeth and aged between 12-25 years were included. The participants were randomly assigned into three groups of 13 each; (1) MI Paste Plus + routine home care; (2) Remin Pro + routine home care; and (3) routine home care (control). The treatment/ observation period was 12 weeks after bracket debonding. Fluorescence loss (∆F, %), lesion area (LA, mm2), lesion volume (∆Q, % × mm2), maximum fluorescence loss (∆Fmax), ICDAS II criteria of WSLs were measured at beginning (T0) and 4 (T1), 8 (T2), and 12 (T3) weeks later. Statistical significance was set at p<0.05.

DETAILED DESCRIPTION:
This randomized controlled trial was a parallel arm 1-1 allocations. The study carried out in the Orthodontics Department, Izmir Katip Celebi University, Turkey. The protocol of the trial was approved by the Izmir Katip Celebi University Research Ethics Committee. A power analysis was carried out to provide that there was enough power to apply a statistical test of the research hypothesis to compare caries regression of Remin Pro to MI Paste Plus comparing with a control group in the remineralization of postorthodontic WSLs. Patients who finished their fixed appliance treatment in the clinic of the Department of Orthodontics, Faculty of Dentistry, Izmir Katip Celebi University who were found to comply with the study criteria were informed. Patients and parents who agreed to participate in the study signed an informed consent. A total of 39 people, 22 women and 17 men, aged between 14 and 23, were included in the study, with 13 people in each group. Gender distribution and average age of the groups are similar. Patients who are 12 to 25 years of age, at least had 12 months of orthodontic treatment with braces, at least had one upper anterior tooth with WSL included in the study. Patient who are smoking, with enamel hypoplasia or fluorosis, with active periodontal disease, with dentin caries, with allergy to casein, with previous bleaching excluded. Simple randomization was performed at the start of the study using a random number table prepared using SPSS software (version 26.0; New York, USA) for the allocation of patients who fulfilled all criteria and were willing to participate in this study. Group I: Patients were instructed to use MI Paste Plus (GC Europe, Leuven, Belgium) according to manufacturers instructions. Group II: Patients were instructed to use (Remin Pro, VOCO , Cuxhaven, Germany) a pea-sized amount of the cream. Group III. Patients (control group) used a 1450 ppm fluoridated tooth paste (Colgate Sensitive Pro-Relief, Colgate-Palmolive, Swidnica, Poland) for conventional tooth brushing and instructed to follow a routine home care. The patients were evaluated at baseline (T0) and every 30 days intervals for 3 months. The primary outcome measures were assessment of mineral loss based on fluorescence loss measurements using QLF. Lesions that scored 1 and 2 according to ICDAS II at debonding were included in the study. The buccal surfaces of the teeth were examined and evaluated by light induced fluorescence intraoral camera QLF-D Biluminator,™ (Inspektor-Pro, Amsterdam, Holland) for capturing fluorescent photographs in accordance with the manufacturer's instructions. Fluorescent images of the patient were evaluated in the 'White Spot Lesion' option of the analysis program (QA2.v.1.27). Following five QLF measurements were performed;

1. Depth of lesion (∆F, %) shows the percentage of loss in fluorescence.
2. Lesion area (LA, mm2) refers to the area covered by the demineralized area on the tooth.
3. Lesion volume (∆Q, % × mm2) is derived from the combination of lesion area and lesion depth and represents the volume of the affected enamel.
4. Maximum fluorescence loss (∆Fmax)is related to depth of lesion and mineral loss. Statistical analysis was performed with IBM® SPSS® (version 26. SPSS Inc., IBM Corporation, NewYork, USA). Descriptive statistics are expressed as number of units (n), percent (%), mean ± standard deviation (x ̅±ss), median (M), minimum (min), maximum (max), and interquartile range (IQR) values. The normal distribution of the data was evaluated with the Shapiro Wilk test of normality. Homogenicity of variances was evaluated with Levene's test.The concordance and differences in the first measurements and the second measurements were evaluated with the intra-class correlation coefficient and the paired samples t test. The ages of the groups were compared with one-way analysis of variance. The ΔF, lesion area and ΔFmax values of the groups in T0, T1, T2 and T3 were compared with two-way analysis of variance in repeated measurements. Bonferroni correction was applied in multiple comparisons. ΔQ, ICDAS II score, and difference values from baseline were compared between groups by Kruskal-Wallis analysis. In case of difference with Kruskal-Wallis analysis, Dunn-Bonferroni test was used for multiple comparisons. For ΔQ, ICDAS II score, Friedman analysis was performed for intragroup timepoint comparisons. Bonferroni correction was applied in multiple comparisons for Friedman analysis. Fisher Exact test was used to compare groups with categorical variables. If the chi-square test result was found to be significant, subgroup analyzes were performed with Bonferroni-corrected two-ratio z-test. Statistical significance level was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 25 years of age,
* at least 12 months of orthodontic treatment with braces,
* at least one upper anterior tooth with WSL.

Exclusion Criteria:

* smoking,
* enamel hypoplasia or fluorosis,
* active periodontal disease,
* dentin caries,
* allergy to casein,
* previous bleaching.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Mineral Content Assessment (ΔF / Depth of lesion) | The patients were evaluated at baseline (T0) and every 30 days intervals for 3 months.
  The buccal surfaces of the teeth were examined and evaluated by light induced fluorescence intraoral camera QLF-D Biluminator,™ (Inspektor-Pro, Amsterdam, Holland) for capturing fluorescent photographs in accordance with the manufacturer's instructions.
Mineral Content Assessment (LA / Lesion area) | The patients were evaluated at baseline (T0) and every 30 days intervals for 3 months.
  The buccal surfaces of the teeth were examined and evaluated by light induced fluorescence intraoral camera QLF-D Biluminator,™ (Inspektor-Pro, Amsterdam, Holland) for capturing fluorescent photographs in accordance with the manufacturer's instructions.
Mineral Content Assessment (∆Q / Lesion volume) | The patients were evaluated at baseline (T0) and every 30 days intervals for 3 months.
  The buccal surfaces of the teeth were examined and evaluated by light induced fluorescence intraoral camera QLF-D Biluminator,™ (Inspektor-Pro, Amsterdam, Holland) for capturing fluorescent photographs in accordance with the manufacturer's instructions.
Mineral Content Assessment (∆Fmax / Maximum fluorescence loss) | The patients were evaluated at baseline (T0) and every 30 days intervals for 3 months.
  The buccal surfaces of the teeth were examined and evaluated by light induced fluorescence intraoral camera QLF-D Biluminator,™ (Inspektor-Pro, Amsterdam, Holland) for capturing fluorescent photographs in accordance with the manufacturer's instructions.

SECONDARY OUTCOMES:
Visual Caries Regression Assessment | The patients were evaluated at baseline (T0) and every 30 days intervals for 3 months.
  ICDAS II scoring

CONTACTS AND LOCATIONS:
Locations (1):
- Sevgi Göl Peynirci, Konak, İzmir, Turkey (Türkiye)